CLINICAL TRIAL: NCT05651087
Title: A Randomized Prospective Clinical Trial to Evaluate Efficacy and Safety of LACUDY for Improving Vaginal Environment Among Breast Cancer Survivals Who Receive Anti-estrogen Therapy
Brief Title: Evaluate Efficacy and Safety of LACUDY for Improving Vaginal Environment in Breast Cancer Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gun Oh Chong (Other)
Responsible Party: Sponsor-Investigator, Gun Oh Chong, professor, Kyungpook National University Chilgok Hospital
Organization: Kyungpook National University Chilgok Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACUDY
Record Dates: First submitted 2022-11-08; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Hormone Receptor-positive Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Breast cancer patient who treated with LACUD
  Interventions: Drug: LACUDY
- Observation (No Intervention): Breast cancer patient who does not treated with LACUD

INTERVENTIONS:
Drug: LACUDY — LACUDY:Insert 2mL twice a week for 4 weeks before going to bed
  Other Names: IC-LC02S2Q2
  Arms: Experimental

SUMMARY:
Adjuvant hormone treatments for early breast cancer are associated with frequent bothersome side effects with major negative impact on patients' quality of life and treatment adherence. Patients most commonly report menopausal symptoms including vaginal dryness, vaginal bleeding, and dyspareunia. Even though previous studies have reported that estrogen topical agent relives these symptoms, non-hormonal therapy should be considered first due to concerns about the role of estrogen in breast cancer development. Therefore, this trial is planned to evaluate the efficacy and safety of LacuD (hyaluronic acid, lactic acid and alginate) in the vaginal environment of breast cancer patients receiving hormone therapy.

DETAILED DESCRIPTION:
* Registered subjects are 1:1 randomized using a random sequencing generator (www.random.org). Experimental group with 30 patients and Control group with 30 patinets.
* In the case of the experimental group, LACUDY 2mL is inserted twice a week for a month before going to bed for 4 weeks.

  * Unpack the product and take it out.
  * Remove the cap by turning it.
  * Fit the nozzle to the end of the syringe and turn it to combine.
  * Hold the syringe with the nozzle facing the vulva, insert it about 5-6 cm into the vagina, and then slowly press the tip of the push rod with patient's thumb to inject all the liquid in the syringe into the vagina.
  * Slowly remove the syringe as the nozzle opens.
  * It is recommended to wear a pad as the injected solution may flow out.
* In the case of the control group, they go about their daily lives without any treatment.
* Both the experimental group and the control group are instructed not to administer intravaginal suppositories or other drugs related to vaginal atrophy and sexual function improvement.
* A total of 2 questionnaires were conducted before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Aged 20 to 60 years diagnosed with breast cancer
3. Receiving anti-hormonal therapy
4. Patients who subjectively complain of vaginal dryness
5. Patients without current psychiatric problems
6. Patients who can understand and respond to the contents of the questionnaire
7. Ability to provide informed consent

Exclusion Criteria:

1. Women under 19 and over 61
2. Pregnant woman
3. In case of recurrence or disease progression
4. Patients without sexual experience
5. Unable to provide informed consent

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change of Vaginal health index | Prior to administration, 1 month after LacuD treatment(2 times in total)
  Female Sexual Function Index (FSFI) Quality of life assessed by Breast Version 4 (FACT-B)

SECONDARY OUTCOMES:
Vaginal microbiome | Prior to administration, 1 month after LacuD treatment(2 times in total)
  Take one cervicovaginal swab sample each